CLINICAL TRIAL: NCT03361995
Title: STEMI Cool Pilot Trial to Assess Cooling as an Adjunctive Therapy to Percutaneous Intervention In Patients With Acute Myocardial Infarction (Phase A)
Brief Title: STEMI Cool Pilot Trial to Assess Cooling as an Adjunctive Therapy to PCI In Patients With Acute MI (Phase A)
Acronym: STEMI Cool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ZOLL Circulation, Inc., USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EDC-2309 Rev 15
Record Dates: First submitted 2017-11-08; First posted 2017-12-05 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Acute Myocardial Infarction
Keywords: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cooling + PCI (Experimental): The subjects will be considered to be enrolled in the Test Arm of the trial when all inclusion and exclusion criteria have been met, the informed consent form has been signed, and randomization to the Test Arm of the trial to allow cooling with the Thermogard XP3 IVTM System before and after PCI.
  Interventions: Device: Cooling Procedure using the ZOLL Thermogard XP3 IVTM System; Device: PCI
- PCI only (Active Comparator): The subjects will be considered to be enrolled in the Control Arm of the trial when all inclusion and exclusion criteria have been met, the informed consent form has been signed, and randomization to the Control Arm of the trial to allow PCI only.
  Interventions: Device: PCI

INTERVENTIONS:
Device: Cooling Procedure using the ZOLL Thermogard XP3 IVTM System — Cooling Procedure with ZOLL Thermogard XP3 IVTM System before and after Percutaneous Coronary Intervention (PCI)
  Arms: Cooling + PCI
Device: PCI — Standard of Care for PCI

SUMMARY:
A Multicenter, Prospective, Randomized-Controlled Trial to Assess Cooling as an Adjunctive Therapy to Percutaneous Intervention In Patients with Acute Myocardial Infarction. The Phase A portion of the trial will include 80 enrollments from up to 15 sites.

DETAILED DESCRIPTION:
The overall objective of this randomized trial is to evaluate the Safety and Efficacy of intravascular cooling using the ZOLL Thermogard XP3 IVTM System, as an adjunctive therapy for patients presenting with acute anterior myocardial infarction and undergoing PCI.

The objective of the Phase A trial is to demonstrate successful incorporation of intravascular cooling into US standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is >= 18 years of age.
2. The patient must have symptoms consistent with AMI (i.e. chest pain, arm pain, etc.) and unresponsive to nitroglycerin, with symptoms beginning greater than 60 minutes but less than 4.5 hours prior to presentation at Hospital.
3. Evidence of Acute Anterior MI with ST-segment elevation of >= 0.2 mV in two or more anterior contiguous precordial leads (V1-V4), as confirmed by ECG at baseline.
4. The patient is eligible for primary PCI.
5. The patient's condition and site workflow allow for the feasibility of implementing the cooling protocol within trial protocol specific requirements.
6. The patient or patient's legal representative is willing to provide written, informed consent to participate in this clinical trial.

Exclusion Criteria:

1. The patient has had a previous myocardial infarction.
2. The patient is experiencing cardiogenic shock, systolic blood pressure [SBP] <100 mmHg, HR>100 bpm and arterial oxygen saturation (pulse oximetry) <= 92% without additional oxygen.
3. The patient has known history of Congestive Heart Failure (CHF), hepatic failure, end stage kidney disease or severe renal failure (clearance < 30ml/min/1.73m²).
4. The patient is presenting with resuscitated cardiac arrest, atrial fibrillation, or Killip risk stratification class III through IV.
5. The patient has an aortic dissection or requires an immediate surgical or procedural intervention other than PCI.
6. The patient is febrile (temperature > 37.5 °C) or has experienced any infection in the last 5 days.
7. The patient has a known previous CABG.
8. The patient has a known recent stroke within 90 days of admission.
9. Cardio-pulmonary decompensation that has occurred en route to the hospital or, in the opinion of the physician, that is imminent or likely to occur following presentation to the clinical site.
10. Contraindications to hypothermia, such as patients with known hematologic dyscrasias which affect thrombosis (e.g., cryoglobulinemia, sickle cell disease, serum cold agglutinins) or vasospastic disorders (such as Raynaud's or thromboangitis obliterans).
11. Any contraindication to cardiac Magnetic Resonance Imaging (MRI), or any implant in the upper body which may cause artifacts on cardiac MRI imaging.
12. The patient has a known hypersensitivity or contraindication to aspirin, heparin, or anaphylaxis to contrast media, which cannot be adequately pre-medicated.
13. The patient has a known history of bleeding diathesis, coagulopathy, cryoglobulinemia or sickle cell anemia, or will refuse blood transfusions.
14. The patient has a height of <1.5 meters (4 feet 11 inches).
15. The patient has a known hypersensitivity or contraindication to Buspirone hydrochloride or Meperidine and/or has been treated with a monoamine oxidase inhibitor in the past 14 days.
16. Patient has a known history of untreated hypothyroidism, Addison's disease, benign prostatic hypertrophy, or urethral stricture that in the opinion of the physician would be incompatible with Meperidine administration.
17. The patient has an Inferior Vena Cava filter in place (IVC).
18. The patient has an anticipated life expectancy of <1 year.
19. The patient has a known, unresolved history of drug use or alcohol dependency, or lacks the ability to comprehend or follow instructions.
20. The patient is currently enrolled in another investigational drug or device trial.
21. The patient is apprehensive about or unwilling to undergo the required MRI imaging at follow-up, has a documented or suspected diagnosis of claustrophobia, or has a Gadolinium allergy.
22. The patient has received thrombolytic therapy en route to the hospital.
23. The patient has received any oral P2Y12 inhibitors prior to enrollment.
24. The patient shows clinical evidence of spontaneous reperfusion as observed symptomatically and/or from ECG findings (partial or complete ST resolution in ECG prior to informed consent and randomization).
25. The patient is a vulnerable subject, for instance, a person in detention (i.e., prisoner or ward of the state).
26. The patient is a female who is known to be pregnant or expected to become pregnant.
27. In the opinion of Investigator or designee the patient is not willing and able to comply with all the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Phase A Safety Endpoint: Incidence of MACE at 30 days. | Through study completion, approximately 1 year
  MACE is defined as Subjects who experienced any of the following events:
  * All-cause death (cardiac, vascular, non-cardiovascular)
  * Myocardial infarction (MI)
  * Clinically-indicated target vessel revascularization (CI TVR)
  * Definite or probable stent thrombosis (ST)
  * New or worsening heart failure (HF) after 24 hours from the end of index PCI, or subsequent re-hospitalization for HF
  * Stroke
  * Major bleeding
Phase A Device Performance Endpoint: Proportion of cooled patients who reach ≤34° at PCI. | Through study completion, approximately 1 year

SECONDARY OUTCOMES:
Phase A Secondary Safety Endpoint 1: Proportion of patients reaching <90 min door-to-balloon time. | Through study completion, approximately 1 year
  The performance goal is at least 93.5% of the patients in Phase A, with Test and Control arms evaluated separately.
Phase A Secondary Safety Endpoint 2: Rate of a composite safety endpoint at 30 days. | Through study completion, approximately 1 year
  Rate of a composite safety endpoint at 30 days defined as the following:
  * Cardiovascular death
  * Myocardial infarction (MI)
  * Clinically-indicated target vessel revascularization (CI TVR)
  * Definite or probable stent thrombosis (ST)
  * New or worsening heart failure (HF) after 24 hours from the end of index PCI, or subsequent re-hospitalization for HF
  * Stroke
  * Major bleeding

IPD SHARING:
Plan to Share IPD: Undecided
The study is registered on ClinicalTrials.gov to make information about the trial publicly available. At all times, including early termination of the study, the sponsors will comply with the reporting requirements of applicable clinical trials registered on ClinicalTrials.gov under the FDA Amendments Act (FDAAA).